CLINICAL TRIAL: NCT04225429
Title: Tazemetostat Expanded Access Program for Adults With Epithelioid Sarcoma
Status: No longer available | Type: Expanded Access
Sponsor: Epizyme, Inc. (Industry)
Responsible Party: Sponsor
Organization: Ipsen (Industry)
Other Study IDs: EZH-801
Record Dates: First submitted 2020-01-08; First posted 2020-01-13 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Epithelioid Sarcoma
Keywords: Epithelioid Sarcoma; Oncology; SMARC-B; loss of INI 1; EZH2; Expanded Access; Compassionate Use
MeSH Terms: conditions — Sarcoma; Neoplasms | interventions — tazemetostat

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Drug: Tazemetostat — 800mg/dose taken orally twice every day.

SUMMARY:
A multicenter, open-label expanded access program to provide access to tazemetostat to Epithelioid Sarcoma (ES) patients in serious need who are otherwise unable to participate in a clinical study or whom access is not available through marketed product in the US.

ELIGIBILITY:
Patients with epithelioid sarcoma (ES) are eligible to enroll in the EAP. The patient with ES must have an advanced disease that is considered life threatening at the time of enrollment and appropriate, comparable, or satisfactory alternative treatments must have been tried without clinical success. Patients with conditions other than ES are not eligible for the tazemetostat EAP.

Inclusion Criteria:

1. Age (at the time of consent): ≥18 years of age.
2. They are unable to participate in tazemetostat clinical trials for their condition.
3. Can provide signed written informed consent.
4. Morphology and immunophenotypic panel consistent with epithelioid sarcoma (e.g., CD34, epithelial embrane antigen [EMA], Keratin, and INI1).
5. Female patients of childbearing potential should:

   * Agree to practice one highly effective method of contraception and one additional effective barrier method (eg, condom or diaphragm with spermicide) at the same time, from the time of providing voluntary written informed consent through 30 days or 5 half-lives (whichever is longer) after the last dose of tazemetostat, and
   * Have a negative beta-human chorionic gonadotropin (β-hCG) pregnancy test at time of screening and within 14 days prior to planned first dose of tazemetostat (urine or serum test is acceptable however, positive urine tests must be confirmed with serum testing), and
   * Agree to use effective contraception from start of screening until 30 days following the last dose of tazemetostat and have a male partner who uses a condom, or
   * Practice true abstinence, (when this is in line with the preferred and usual lifestyle of the patient) or
   * Have a male partner who is vasectomized.
6. Male patients with a female partner of childbearing potential should:

   * Be vasectomized, or
   * Agree to use condoms from at least 7 days prior to initiating and during tazemetostat treatment and for at least 30 days following the last dose of tazemetostat, or
   * Have a female partner who is NOT of childbearing potential.

Exclusion Criteria:

* 1. Is unwilling to exclude grapefruit juice, Seville oranges and grapefruit from the diet and all foods that contain those fruits from time of enrollment while on the EAP.

  2. Is currently taking any prohibited medication(s) as described in Section 6.3 of the protocol.

  3. Has known hypersensitivity to any of the components of tazemetostat or other inhibitor(s) of EZH2.

  4. Has thrombocytopenia, neutropenia, or anemia of Grade ≥3 (per CTCAE v5.0 criteria) within the past month, or any prior history of myeloid malignancies, including myelodysplastic syndrome (MDS).

  5. Is known to have any abnormalities associated with MDS (e.g. del 5q, chr 7 abn) and MPN (e.g. JAK2 V617F) observed in cytogenetic testing and DNA sequencing.

  6. Has a prior history of T-LBL/T-ALL. 7. For female patients of childbearing potential: Is pregnant or nursing. 8. For male patients: Is unwilling to adhere to contraception criteria from at least 7 days prior to initiating and during tazemetostat treatment and for at least 30 days after last dose of tazemetostat.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen